CLINICAL TRIAL: NCT04658511
Title: Correlation Between the Presence of the Arcade of Struthers on Preoperative Ultrasound and During Endoscopic Surgery
Brief Title: Presence of the Arcade of Struthers on Preoperative Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Collaborators: Kleinert, Kutz and Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20.1097
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Cubital Tunnel Syndrome
Keywords: arcade of struthers; cubital tunnel
MeSH Terms: conditions — Cubital Tunnel Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants (Experimental): Patients diagnosed with cubital tunnel syndrome who are being scheduled for a primary endoscopic cubital tunnel release by the principle investigator will be recruited
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — On the spot, during the pre-op clinic visit, an ultrasound exam will be done by the PI trying to visualize the arcade of Struthers

SUMMARY:
To determine the correlation between the presence of the arcade of Struthers on preoperative ultrasound and during endoscopic surgery for cubital tunnel syndrome, and to determine the reliability of a portable ultrasound probe to detect the arcade of Struthers in the arm.

DETAILED DESCRIPTION:
The ulnar nerve comes from the medical cord of the brachial plexus (C8-T1). It travels out of the axilla along the medial border of the arm to pass into the forearm via the cubital tunnel at the elbow. Cubital tunnel syndrome is the result of compression and traction on the ulnar nerve about the elbow, which can occur at multiple sites. The most proximal possible site of compression causing is the arcade of Struthers. This entity has been described as an aponeurotic band, as a fibrous canal or as thickened connective tissue. Regardless of the nomenclature, ulnar nerve compression has been documented at the location of the arcade of Struthers, which is 6 to 10 cm proximal to the medial epicondyle. Simple open in situ decompression typically results in decompression of the ulnar nerve 6 cm proximal and 6 cm distal to the medial epicondyle while endoscopic ulnar nerve decompression decompresses on average 17 cm of the ulnar nerve (range 25-23 cm), thus consistently reaching the area of the arcade of Struthers. Recurrent cubital tunnel syndrome after simple decompression can be due failure to the release of the arcade of Struthers, and the revision surgery involved extending the incision and length of ulnar nerve release. With the advances in ultrasound imaging, the identification of the arcade of Struthers in mid arm is feasible. hence, it would be beneficial to identify the presence and the location of the arcade of Struthers pre-operatively, to direct the surgical procedure to decompress the ulnar nerve more proximally in cases of a simple decompression in situ.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cubital tunnel syndrome
* Planned for endoscopic cubital tunnel release primary surgery
* >=18 years of age
* no previous arm or elbow surgeries

Exclusion Criteria:

* Revision surgery
* Planned for open cubital tunnel release
* Prior surgical intervention around the arm or the elbow
* <18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Presence of the arcade of Struthers | through study completion, average of 1 day/visit
  Presence/visualization of the arcade of Struthers with ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Tuna Ozyurekoglu, MD, Principal Investigator — President, Christine M Kleinert Institute for Hand and Microsurgery
Locations (2):
- United States (2):
  - Christine M Kleinert Institute, Louisville, Kentucky
  - Kleinert Kutz & Associates, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No
No plan to share with other researchers

REFERENCES:
- [Result] Andrews K, Rowland A, Pranjal A, Ebraheim N. Cubital tunnel syndrome: Anatomy, clinical presentation, and management. J Orthop. 2018 Aug 16;15(3):832-836. doi: 10.1016/j.jor.2018.08.010. eCollection 2018 Sep. PMID 30140129
- [Result] Staples JR, Calfee R. Cubital Tunnel Syndrome: Current Concepts. J Am Acad Orthop Surg. 2017 Oct;25(10):e215-e224. doi: 10.5435/JAAOS-D-15-00261. PMID 28953087